CLINICAL TRIAL: NCT02552043
Title: Video Game Exercise Effectiveness of a Domiciliary Pulmonary Rehabilitation Program in Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Tamara del Corral Núñez-Flores, Msc, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAMadrid
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Exercise capacity; Interactive gaming console; Pulmonary rehabilitation
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nintendo Wii exercise program group (Experimental): The EG will perform a domiciliary Pulmonary Rehabilitation program of 30-60 min exercise, 5 days/week during 6 weeks using a Nintendo Wii platform with the game EA SPORTS ACTIVE 2. The exercise activities were loaded into each participant´s console during the clinical interview and adjusting the exercises according to their age in 2 groups (>12 years and <13 years). The program consisted of 6 different workouts (1st and 2nd weeks: legs exercises; 3rd week: upper limb exercises; 4th week: thorax exercises; 5th and 6th weeks: cardio exercises), so the patients had a gradual increase reaching the maximum load at the end of training.
  Interventions: Other: Nintendo Wii exercise program
- Control group (No Intervention): The CG carried out their routine patient management

INTERVENTIONS:
Other: Nintendo Wii exercise program — The aerobic training protocol was designed to improve muscular strength, body endurance and flexibility (involved activities as: running, up the knees, butt kickers, etc.). The game used has a strap pouch to hold the Nunchuk© controller placed on the thigh that detects the lower body movements, and also features a number of exercise options supervised by a virtual personal trainer
  Arms: Nintendo Wii exercise program group

SUMMARY:
The aim of this study is to evaluate the efficacy of a long-term domiciliary exercise program using the Wii video game platform as a training modality in Cystic Fibrosis (CF) patients. Investigators hypothesize that an exercise program performed by active videogames (AVG) will produce an improvement in exercise tolerance and muscular strength to be maintained over time in young CF patients.

DETAILED DESCRIPTION:
This is a randomized and longitudinal trial. Participants will be randomize in 2 groups: control group (CG) and experimental group (EG), by the ©GrapfPad Software, Inc. The CG will carry out their routine patient management, and the EG will perform also a domiciliary Pulmonary Rehabilitation program of 30-60 min exercise, 5 days/week during 6 weeks using a Nintendo WiiTM platform with the game EA SPORTS ACTIVE 2.

Before and after we will measure:

1. exercise tolerance using the six minutes walk test (6MWT) and the modified shuttle walk test (MSWT);
2. muscular strength using horizontal jump test (HJT), medicine ball throw (MBT) and handgrip strength (right hand (HGR); left hand (HGL)); and
3. HRQoL using the 3 versions of the Cystic Fibrosis Questionnaire-Revised (CFQ-R 6-11, CFQ-R 14+, CFQ-R Parents).

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of CF, clinically stable without exacerbations of the disease in the previous 6 weeks to the inclusion date.

Exclusion Criteria:

* To present clinical evidence of cardiovascular, neuromuscular or osteo-articular comorbidities that limit the participation in exercise programs.
* Lung transplant candidates and those patients that followed any kind of rehabilitation program 12 months before the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The six-minute walk test (6MWT) | Change from Baseline in the 6-min walk distance at 6 weeks and at 12 months of follow up period
  The six-minute walk test (6MWT) will perform following the American Thoracic Society recommendations. It is a valid and reliable test in CF children. After recorded basal measurements, patients will be asked to walk as much as possible and standardized encouragement will be given after each minute. Two tests will be performed and the highest walking distance will be recorded.
The modified shuttle walk test (MSWT) | Change from Baseline in the modified shuttle walk distance at 6 weeks and at 12 months of follow up period
  The modified shuttle walk test (MSWT): consisted of 15 levels in which patients should walk quickly, gradually increasing speed on a 10 meters space. An external audio signal indicates a level shift. Two tests were performed with 30 minutes of rest and the highest walking distance was recorded (MSWD). Valid and reliable test to measure exercise tolerance in CF.

SECONDARY OUTCOMES:
Horizontal jump test (HJT) | Change from Baseline in the horizontal jump distance at 6 weeks and at 12 months of follow up period
  Horizontal jump test (HJT): was made with feet placed at shoulder height. Jump would be invalid if they give an extra step and if they are unbalanced and touch the floor with their hands. Three jumps were made and the highest distance in centimetres was recorded. Horizontal jump assessment is has shown reliable to evaluate the power of the legs.
Medicine ball throw (MBT) | Change from Baseline in the throw distance at 6 weeks and at 12 months of follow up period
  Medicine ball throw (MBT): was performed sitting on their knees before throwing the medicine ball (<12 years 2kg; >13 years 3kg) forward like a chest pass with both hands. The furthest distance of the three throws was recorded, with a 1-2 minutes rest between each throw. This instrument is valid and reliable for kindergarten children.
Handgrip strength (HG) | Change from Baseline in handgrip isometric strength at 6 weeks and at 12 months of follow up period
  Handgrip strength will be calculate using a Hand Dynamometer (Jamar® hydraulic USA) of 90Kg. Three trails will given for each hand separately with 30s rest between them and the highest value was recorded in kg (right hand (HGR); left hand (HGL)). The subject is placed sitting with the dynamometer in an angle of 90°. This device is valid and reliable to measure isometric strength and anaerobic endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Superior de estudios Universitarios La SALLE, Aravaca, Madrid, Spain